CLINICAL TRIAL: NCT01024582
Title: Image Guided Preoperative Accelerated Partial Breast Irradiation (PAPBI): Defining Radiotherapy Sensitivity
Brief Title: Radiation Therapy Followed by Surgery in Treating Patients With Early-Stage Breast Cancer
Acronym: PAPBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M08PBI; NL24996.031.08 (Registry Identifier: CCMO); EU-20989
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; invasive breast cancer; adenocarcinoma of the breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy; Biopsy, Fine-Needle; Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- accelerated partial breast irradiation (Experimental): pre-operative radiation of the in situ tumor in the breast
  Interventions: Procedure: biopsy; Procedure: fine-needle aspiration; Radiation: accelerated partial breast irradiation; Radiation: image-guided radiation therapy

INTERVENTIONS:
Procedure: biopsy — before treatment a biopsy will be taken to confirm breast cancer type
Procedure: fine-needle aspiration — at FNA tumor material will be collected and fresh frozen for micro-analyses; parafin embedded tissue will bestored for tissue-array analysis
Radiation: accelerated partial breast irradiation
Radiation: image-guided radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving CT-guided accelerated radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This clinical trial is studying giving radiation therapy followed by surgery to see how well it works in treating patients with early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* is to investigate the impact of a short fractionated schedule given preoperatively on local control, cosmesis and breast fibrosis.
* To further design optimal treatment strategies for individual breast cancer patients treated with breast-conserving therapy (BCT) on the basis of biological parameters, including the expression profile of the primary tumor, for both m-RNA as for micro-RNA, with first, a focus on radiotherapy responsiveness and second, on local recurrence rate, distant metastases and survival.
* proteomics will be studied in fine-needle aspiration samples. A classifier can be build (genomic or proteomic or any kind of molecular signature) to identify responders and non-responders
* quality of life

OUTLINE: Patients undergo image-guided preoperative accelerated partial-breast irradiation (PAPBI) 10 times over 12 days (10 x 4 Gy) and later in the study 5 times 6 Gy. Six weeks after completion of image-guided PAPBI, patients undergo surgery.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of unifocal cT1-2 (1-3 cm) pN0 M0 breast cancer
* Must have undergone a sentinel node procedure prior to irradiation

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2009-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
local recurrence | 5 years
  Local recurrences should not exceed 4% at 5 years of follow-up

SECONDARY OUTCOMES:
breast fibrosis | 5 years
  decrease from 27% as found in the boost arm of the EORTC boost-no boost trial to 15%
cosmetic outcome | 5 years
  is anticipated that the overall score for cosmetic outcome will be superior compared to conventional whole breast postoperative radiotherapy plus boost.
Pathological response | 6 weeks after finishing iradiation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paula Elkhuizen, MD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Leij F, Bosma SC, van de Vijver MJ, Wesseling J, Vreeswijk S, Rivera S, Bourgier C, Garbay JR, Foukakis T, Lekberg T, van den Bongard DH, van Vliet-Vroegindeweij C, Bartelink H, Rutgers EJ, Elkhuizen PH. First results of the preoperative accelerated partial breast irradiation (PAPBI) trial. Radiother Oncol. 2015 Mar;114(3):322-7. doi: 10.1016/j.radonc.2015.02.002. Epub 2015 Feb 17. PMID 25701298